CLINICAL TRIAL: NCT06232941
Title: Comparative Evaluation of Three Calcium Silicate Based Materials as Pulpotomy Agents for Permanent Mature Molars With Irreversible Pulpitis: Randomized Clinical Trial
Brief Title: Comparative Evaluation of Three Pulpotomy Agents for Permanent Mature Molars With Irreversible Pulpitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-REC1261
Record Dates: First submitted 2023-09-13; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-09

CONDITIONS: Vital Pulp Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Odontocem pulpotomy agent (Experimental): calcium silicate-based technology containing 0.2% of the low steroid triamcinolone acetonide and has outstanding biocompatibility, handling properties and least amount of staining potential
  Interventions: Procedure: Full pulpotomy procedure
- NeoPutty bioceramic (Active Comparator): premixed format of tricalcium silicate-based material (Bioceramic). It's composed of tantalum oxide, tricalcium silicate, calcium aluminate, dicalcium silicate, tricalcium aluminate, and calcium sulfate
  Interventions: Procedure: Full pulpotomy procedure
- Mineral Trioxide Aggregate material (Active Comparator): hydrophilic and biocompatible endodontic biomaterial, capable of stimulating healing and osteogenesis
  Interventions: Procedure: Full pulpotomy procedure

INTERVENTIONS:
Procedure: Full pulpotomy procedure — vital pulp therapy for molars with irreversible pulpitis instead of doing root canal treatment
  Other Names: vital pulp therapy

SUMMARY:
Statement of the problem:

Accurate pulpal diagnosis is essential for decision making between vital pulp therapy and root canal treatment. Clinical and radiographic examinations do not correctly reflect the histological state of the pulp and consequently its ability to heal. Also, despite the various advantages of using MTA as a pulp capping agent, it has several drawbacks.

Aim of the study:

The aim of the study is to compare two types of calcium silicate-based materials to MTA in permanent mature molars diagnosed with irreversible pulpitis regarding the following parameters; level of inflammatory biomarker level, clinical and radiographic outcomes.

Materials and methods:

Thirty-six patients with mature permanent molars exhibiting signs and symptoms indicative of irreversible pulpitis will be enrolled. A careful periodontal treatment and standardized operative procedure will be followed for all participants. Gingival crevicular fluid samples will be obtained before any local anesthetics' administration, followed by isolation of teeth with a dental dam and removal of caries. Pulpotomy will be performed using sterile round bur till level of orifices and then haemostasis will be achieved using sodium hypochlorite. At this point, patients will be randomly divided into three groups of 12 depending on the type of calcium silicate-based material used. Later, resin modified glass ionomer will be applied, etching, bonding and placement of composite as the permanent restoration. Follow up clinically and radiographically will be done.

DETAILED DESCRIPTION:
For many centuries, there has been a closely held belief that any vital mature permanent tooth diagnosed with irreversible pulpitis will require root canal treatment. The reason for such treatment modality, is the high success rate reaching 100% if performed with high standards(1). However, many studies have demonstrated that root canal therapy can be time-consuming(2), necessitate multiple visits(3), be expensive for both the patient and the dentist, and can increase the likelihood that the tooth will fracture because of the loss of tooth structure(2).

On the other hand, vital pulp therapy (VPT) provides many advantages compared to root canal treatment. For example; it maintains the proprioceptive sensation of the tooth, biological immune response from the retained pulp tissue can prevent infection of the apical area, regenerative and repair potential of the pulp is retained, structural integrity of the tooth is maintained, lowering the risk of fracture and there is a notable decrease in pain and discomfort for the patient (4).

More conservative VPT like pulpotomy was limited to immature teeth with mechanical, carious, or traumatic pulp exposure who don't exhibit any periapical disease. In such cases, the goal has been to ensure completion of root formation (apexogenesis)(5). However, the European Society of Endodontology (ESE) and the American Association of Endodontists (AAE) recently released position statements stating that "pre-treatment diagnosis of irreversible pulpitis is not necessarily an indication for pulpectomy", ushering in a new era for minimally invasive VPT in mature permanent teeth Although, several studies (8,14)found that using mineral trioxide aggregate (MTA) for VPT of cariously exposed permanent teeth with irreversible pulpitis resulted in high clinical success rates. Clinically, there have been various complaints against MTA. There have been reports of difficult handling, prolonged setting time, expensive cost, and probable tooth discoloration By far, the most popular and widely utilized materials in the endodontic therapy are calcium silicate cements. Odontocem (Australian Dental Manufacturing, Brisbane, Australia) is a calcium silicate-based technology containing 0.2% of the low steroid triamcinolone acetonide and has outstanding biocompatibility, handling properties and least amount of staining potential. It can be utilised as a dentine substitute for lining deep cavities. Odontocem is proposed to provide antibacterial activity due to its initial high PH and pain relief due to the presence of a potent steroid (16).

Another calcium silicate material that is also recently introduced in the market is NeoPutty (Avalon Biomed Inc., Bradenton, USA). NeoPutty is premixed format of tricalcium silicate-based material (Bioceramic). It's composed of tantalum oxide, tricalcium silicate, calcium aluminate, dicalcium silicate, tricalcium aluminate, and calcium sulfate(17). Guillen et al 2022 (17)compared the cytocompatibility of NeoPutty to NeoMTA Plus and MTA Angelus and concluded that all three materials provided adequate cytocompatibility and preliminary evidence that NeoPutty can be used as pulp capping agent in VPT.

ELIGIBILITY:
Inclusion Criteria:

* Participants with permanent molars considered as having clinical signs and symptoms consistent with a diagnosis of irreversible pulpitis if they presented with the following chief complaint:
* Intermittent or spontaneous, sharp or dull, localized, diffuse, or referred pain.
* Rapid exposure to dramatic temperature changes elicited heightened and --prolonged episodes of pain even after the thermal stimulus has been removed.
* Participants without signs and symptoms of apical periodontitis
* Periodontally healthy permanent molars
* Systemically healthy patients without any history of long-acting NSAIDs intake in the past one week will be included to eliminate any confounding factors.

Exclusion Criteria:

* Non-restorable teeth with cracks or subgingival caries, associated sinus or swelling, immature roots, periapical rarefaction (PAI score ≥ 3).
* Poor periodontal support.
* Negative response to pulp sensibility tests.
* Diabetic, immune-compromised, pregnant patients
* Patient had a positive history of antibiotic use in the past 1 month or required antibiotic prophylaxis
* The tooth was previously accessed
* The tooth had an inflamed pulp in which bleeding could not be controlled within 10 minutes.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Inflammatory marker level (matrix metalloproteinase 9) for assessment of pulpotomy success. | Inflammatory biomarker level in gingival crevicular fluid using ELISA kit at the day of the procedure and then after 1 week .
  Inflammation biomarker which is matrix metalloproteinase 9 (diagnostic) may be provided by molecules expressed during the cascade of tissue inflammation. Also, studies have demonstrated that the presence of protein markers or biomarkers in gingival crevicular fluid (GCF) can represent pulpal events

SECONDARY OUTCOMES:
Radiographic evaluation | baseline, after 6 and 12 months
  Using CBCT, periapical index scale will be used to assess presence or absence of radiolucency associated with the tested teeth Radiographically (baseline, -6 and -12 months) concerning any changes in tooth and surrounding structures.

IPD SHARING:
Plan to Share IPD: No